CLINICAL TRIAL: NCT02088554
Title: Medtronic PERIcardial SurGical AOrtic Valve ReplacemeNt Pivotal Trial A Multi-center, Non-randomized Trial to Determine the Safety and Effectiveness of the Model 400 Aortic Valve Bioprosthesis in Patients With Aortic Valve Disease
Brief Title: PERIGON Pivotal Trial
Acronym: PERIGON
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Surgery (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PERIGON
Record Dates: First submitted 2014-03-04; First posted 2014-03-17 (Estimated); Results first posted 2024-06-04 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Model 400 aortic valve bioprosthesis (Experimental)
  Interventions: Device: Model 400 aortic valve bioprosthesis

INTERVENTIONS:
Device: Model 400 aortic valve bioprosthesis

SUMMARY:
To evaluate the safety and effectiveness of the Model 400 aortic valve bioprosthesis.

DETAILED DESCRIPTION:
This is a prospective, interventional, non-randomized, worldwide, multi-center trial. A maximum of 1300 subjects were to be implanted at a maximum of 40 sites in the US, Europe and Canada. The trial includes male and female patients of legal age to provide informed consent in the country where they enrolled in the trial, requiring replacement for a diseased, damaged, or malfunctioning native or prosthetic aortic valve. Subjects are followed out to 5 years, and select sites follow subjects out to 12 years. Enrollment closed on 14Jul2017 for all valve sizes. Enrollment was reopened in Apr2019 for the 29mm valve size at a subset of US and Canadian sites to obtain greater patient numbers required by the FDA to support US commercial approval of this valve size. Enrollment for the 29mm valve size closed on 14Feb2023.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has moderate or greater aortic stenosis or regurgitation, and there is clinical indication for replacement of their native or prosthetic aortic valve with a bioprosthesis, with or without concomitant procedures, which are limited to any of the following:

   i. Left atrial appendage (LAA) ligation ii. CABG (coronary artery bypass grafting) iii. Patent foramen ovale (PFO) closure iv. Ascending aortic aneurysm or dissection repair not requiring circulatory arrest v. Resection of a sub-aortic membrane not requiring myectomy
2. Patient is geographically stable and willing to return to the implanting site for all follow-up visits
3. Patient is of legal age to provide informed consent in the country where they enroll in the trial
4. Patient has been adequately informed of risks and requirements of the trial and is willing and able to provide informed consent for participation in the clinical trial

Exclusion Criteria:

1. Patient has a pre-existing prosthetic valve or annuloplasty device in another position or requires replacement or repair of the mitral, pulmonary or tricuspid valve
2. Patient has had previous implant and then explant of the Model 400 aortic valve bioprosthesis
3. Patient presents with active endocarditis, active myocarditis or other systemic infection
4. Patient has an anatomical abnormality which would increase surgical risk of morbidity or mortality, including:

   * Ascending aortic aneurysm or dissection repair requiring circulatory arrest
   * Acute Type A aortic dissection
   * Ventricular aneurysm
   * Porcelain aorta
   * Hostile mediastinum
   * Hypertrophic obstructive cardiomyopathy (HOCM)
   * Documented pulmonary hypertension (systolic >60mmHg)
5. Patient has a non-cardiac major or progressive disease, with a life expectancy of less than 2 years. These conditions include, but are not limited to:

   * Child-Pugh Class C liver disease
   * Terminal cancer
   * End-stage lung disease
6. Patient has renal failure, defined as dialysis therapy or glomerular filtration rate(GFR)<30 mL/min/1.73 m2
7. Patient has hyperparathyroidism
8. Patient is participating in another investigational device or drug trial or observational competitive study
9. Patient is pregnant, lactating or planning to become pregnant during the trial period
10. Patient has a documented history of substance (drug or alcohol) abuse
11. Patient has greater than mild mitral valve regurgitation or greater than mild tricuspid valve regurgitation as assessed by echocardiography
12. Patient has systolic ejection fraction (EF)<20% as assessed by echocardiography
13. Patient has Grade IV Diastolic Dysfunction
14. Patient has documented bleeding diatheses
15. Patient has had an acute preoperative neurological deficit or myocardial infarction and has not returned to baseline or stabilized ≥30 days prior to enrollment
16. Patient requires emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1312 (Actual)
Dates: Start 2014-05-12 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2035-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sabik, MD, Principal Investigator — University Hospital Cleveland Medical Center (Not a recruiting site); Prof. Dr. Robert Johannes Menno Klautz, MD, Principal Investigator — Leiden University Medical Center
Locations (38):
- United States (20):
  - University of Southern California (USC) University Hospital, Los Angeles, California
  - University of Colorado Hospital, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - University of Florida Shands, Gainesville, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Cardiovascular Center, Ann Arbor, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Maimonides Medical Center, Brooklyn, New York
  - The Mount Sinai Medical Center, New York, New York
  - New York-Presbyterian Hospital/Columbia University Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Riverside Methodist Hospital (OhioHealth), Columbus, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Cardiothoracic and Vascular Surgeons (CTVS), Austin, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
- Canada (5):
  - London Health Sciences Centre - University Campus, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec
  - Toronto General Hospital, Toronto
- France (2):
  - Hôpital Cardiologique du Haut-Lévêque, Bordeaux
  - Hôpital Bichat - Claude Bernard, Paris
- Germany (5):
  - Uniklinik Köln, Cologne, Köln
  - Deutsches Herzzentrum München, Munich, München
  - Universitäts Klinikum Frankfurt - Goethe-Universität, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Herzzentrum Leipzig GmbH, Leipzig
- Ospedale San Raffaele - Milano, Milan, Italy
- Netherlands (2):
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Erasmus MC, Rotterdam
- Switzerland (2):
  - Inselspital - Universitätsspital Bern, Bern
  - UniversitätsSpital Zürich, Zurich
- Guy's & St Thomas' NHS Foundation Trust - St Thomas' Hospital, London, United Kingdom

REFERENCES:
- [Derived] Velders BJJ, Vriesendorp MD, Weissman NJ, Sabik JF 3rd, Reardon MJ, Dagenais F, Moront MG, Rao V, Fukuhara S, Gunzinger R, van Leeuwen WJ, Brown WM, Groenwold RHH, Klautz RJM, Asch FM. Core Laboratory Versus Center-Reported Echocardiographic Assessment of the Native and Bioprosthetic Aortic Valve. Echocardiography. 2024 Dec;41(12):e70047. doi: 10.1111/echo.70047. PMID 39624936
- [Derived] Klautz RJM, Rao V, Reardon MJ, Deeb GM, Dagenais F, Moront MG, Little SH, Labrousse L, Patel HJ, Ito S, Li S, Sabik JF 3rd, Oh JK. Examining the typical hemodynamic performance of nearly 3000 modern surgical aortic bioprostheses. Eur J Cardiothorac Surg. 2024 May 3;65(5):ezae122. doi: 10.1093/ejcts/ezae122. PMID 38710669
- [Derived] Velders BJJ, Vriesendorp MD, De Lind Van Wijngaarden RAF, Rao V, Reardon MJ, Shrestha M, Chu MWA, Sabik JF 3rd, Liu F, Klautz RJM. Perioperative care differences of surgical aortic valve replacement between North America and Europe. Heart. 2023 Jun 26;109(14):1106-1112. doi: 10.1136/heartjnl-2023-322350. PMID 36963820
- [Derived] Klautz RJM, Kappetein AP, Lange R, Dagenais F, Labrousse L, Bapat V, Moront M, Misfeld M, Zeng C, Sabik Iii JF; PERIGON Investigators. Safety, effectiveness and haemodynamic performance of a new stented aortic valve bioprosthesis. Eur J Cardiothorac Surg. 2017 Sep 1;52(3):425-431. doi: 10.1093/ejcts/ezx066. PMID 28475690

RESULTS

PARTICIPANT FLOW:
Groups:
- Medtronic Model 400 Avalus Bioprosthetic Aortic Valve: The Medtronic Model 400 Avalus Bioprosthetic Aortic Valve is indicated for patients who require replacement of their native aortic valve.
Period: Overall Study
Arm/Group | Medtronic Model 400 Avalus Bioprosthetic Aortic Valve
Started | 1312
Implanted | 1132
1 Year Completion (Primary outcome milestone (a minimum of 15 participants per valve size completes 1 year follow-up)) | 1050
Completed (Participants who have completed 5 year follow-up) | 268
Not Completed | 1044
Not completed — Exited before procedure | 130
Not completed — Attempted but not implanted | 31
Not completed — Implant not attempted | 19
Not completed — Pending next visit | 532
Not completed — Death | 170
Not completed — Subject Withdrew + Physician Withdrew + Subject Not Implanted With Study Valve | 96
Not completed — Lost to Follow-up | 23
Not completed — Explanted | 32
Not completed — Any other reason not covered by previous categories | 11

BASELINE CHARACTERISTICS:
Groups:
- Medtronic Model 400 Avalus Bioprosthetic Aortic Valve: Participants implanted with the Medtronic Model 400 Avalus Bioprosthetic Aortic Valve, as indicated for patients who require replacement of their native aortic valve.
Arm/Group | Medtronic Model 400 Avalus Bioprosthetic Aortic Valve
Number analyzed (Participants) | 1132
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 278
  Male | 854
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 638
  Unknown or Not Reported | 475
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 636
  More than one race | 0
  Unknown or Not Reported | 476
Region of Enrollment [Number; unit: participants]
  Canada | 268
  Europe | 475
  United States | 389
New York Heart Association (NYHA) Classification [Count of Participants; unit: Participants] — Measure of heart failure severity (lower class desirable) I - No limitation of physical activity. Ordinary physical activity does not cause fatigue, palpitation or shortness of breath.
  II - Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  III - Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  IV - Symptoms of heart failure at rest. Any physical activity causes further discomfort.
  Participants
    NYHA Class I | 126
    NYHA Class II | 533
    NYHA Class III | 451
    NYHA Class IV | 22

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Safety of the Model 400 Avalus Valve With Regard to Valve-related Adverse Events and Death at 1 Year Post-implant
Description: Safety of the valve is evaluated by the time-related incidence of valve-related adverse events and death. The following valve-related adverse events are evaluated in this study: Thromboembolism, Thrombosis, Hemorrhage, Paravalvular leak (PVL), Endocarditis, Hemolysis, Structural valve deterioration, Non-structural dysfunction, Reintervention, Explant, and Death. A minimum of 15 participants per valve size are evaluated. The incidence rates will be used to summarize valve-related adverse events and death.
Time Frame: 1 year post-implant
Measure: Number; unit: percentage of participants with event
Groups:
- Medtronic Avalus Valve 19mm: Safety evaluation for participants implanted with the 19mm Medtronic Avalus Valve
- Medtronic Avalus Valve 21mm: Safety evaluation for participants implanted with the 21mm Medtronic Avalus Valve
- Medtronic Avalus Valve 23mm: Safety evaluation for participants implanted with the 23mm Medtronic Avalus Valve
- Medtronic Avalus Valve 25mm: Safety evaluation for participants implanted with the 25mm Medtronic Avalus Valve
- Medtronic Avalus Valve 27mm: Safety evaluation for participants implanted with the 27mm Medtronic Avalus Valve
- Medtronic Avalus Valve 29mm: Safety evaluation for participants implanted with the 29mm Medtronic Avalus Valve
- Medtronic Avalus Valve (17mm - 29mm): Safety evaluation for participants implanted with the with Medtronic Avalus Valves sized 17mm - 29mm. One subject implanted with 17mm Avalus Valve included only in composite results to protect privacy.
Arm/Group | Medtronic Avalus Valve 19mm | Medtronic Avalus Valve 21mm | Medtronic Avalus Valve 23mm | Medtronic Avalus Valve 25mm | Medtronic Avalus Valve 27mm | Medtronic Avalus Valve 29mm | Medtronic Avalus Valve (17mm - 29mm)
Number analyzed (Participants) | 42 | 211 | 401 | 350 | 101 | 26 | 1132
percentage of participants with event
  All death | 9.5 | 2.8 | 2.2 | 2.9 | 4.0 | 3.8 | 3.0
  Valve- related death | 0.0 | 0.9 | 0.2 | 0.0 | 0.0 | 0.0 | 0.3
  Thromboembolism | 0.0 | 2.8 | 2.7 | 2.9 | 4.0 | 3.8 | 2.8
  Valve thrombosis | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  All hemorrhage | 7.1 | 3.8 | 6.7 | 4.3 | 7.9 | 0.0 | 5.4
  Major hemorrhage | 7.1 | 0.5 | 5.0 | 3.4 | 5.0 | 0.0 | 3.6
  All paravalvular leak | 0.0 | 0.5 | 0.5 | 0.6 | 1.0 | 0.0 | 0.5
  Major paravalvular leak | 0.0 | 0.5 | 0.0 | 0.3 | 0.0 | 0.0 | 0.2
  Endocarditis | 0.0 | 0.5 | 1.5 | 1.4 | 1.0 | 0.0 | 1.1
  Hemolysis | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Non-structural valve dysfunction | 0.0 | 0.5 | 0.5 | 0.6 | 1.0 | 0.0 | 0.5
  Structural valve deterioration | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Severe hemodynamic dysfunction - indeterminate or evolving cause | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Reintervention | 0.0 | 0.9 | 1.2 | 0.6 | 1.0 | 0.0 | 0.9
  Explant | 0.0 | 0.9 | 1.2 | 0.6 | 1.0 | 0.0 | 0.9

2. Primary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to the Change of New York Heart Association (NYHA) Classification From Baseline Through 1 Year
Description: At each timepoint, a minimum of 15 participants per valve size evaluated for change in New York Heart Association (NYHA) functional classification from baseline to 1 year post-procedure.
  Measure Description: Cardiac Disease with Functional Classes (lower value is more desirable than higher value) I - No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  II - Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  III - Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  IV - Symptoms of heart failure at rest. Any physical activity causes further discomfort.
Time Frame: Discharge (up to 30 days), 3-6 months, and 1 year post-implant
Population: Difference in the overall number of participants analyzed and of those analyzed at each timepoint is due to classification not assessed, classification was unable to be assessed, or the participant exited the trial before that timepoint. For 29mm participants, difference in total number of participants analyzed was also due to participants who have not yet reached specified timepoint.
Measure: Count of Participants; unit: Participants
Groups:
- Medtronic Avalus Valve 19mm: Effectiveness evaluation for participants implanted with the 19mm Medtronic Avalus Valve
- Medtronic Avalus Valve 21mm: Effectiveness evaluation for participants implanted with the 21mm Medtronic Avalus Valve
- Medtronic Avalus Valve 23mm: Effectiveness evaluation for participants implanted with the 23mm Medtronic Avalus Valve
- Medtronic Avalus Valve 25mm: Effectiveness evaluation for participants implanted with the 25mm Medtronic Avalus Valve
- Medtronic Avalus Valve 27mm: Effectiveness evaluation for participants implanted with the 27mm Medtronic Avalus Valve
- Medtronic Avalus Valve 29mm: Effectiveness evaluation for participants implanted with the 29mm Medtronic Avalus Valve
- Medtronic Avalus Valve (17mm - 29mm): Effectiveness evaluation for participants implanted with the with Medtronic Avalus Valves sized 17mm - 29mm. One subject implanted with 17mm Avalus Valve included only in composite results to protect privacy.
Arm/Group | Medtronic Avalus Valve 19mm | Medtronic Avalus Valve 21mm | Medtronic Avalus Valve 23mm | Medtronic Avalus Valve 25mm | Medtronic Avalus Valve 27mm | Medtronic Avalus Valve 29mm | Medtronic Avalus Valve (17mm - 29mm)
Number analyzed (Participants) | 42 | 211 | 401 | 350 | 101 | 26 | 1132
Participants
  Discharge up to 30 days: number analyzed (Participants) | 38 | 174 | 302 | 272 | 70 | 23 | 880
  Discharge up to 30 days: Improved 3 Classes | 0 | 0 | 5 | 2 | 2 | 0 | 9
  Discharge up to 30 days: Worsened 1 Class | 0 | 15 | 16 | 18 | 10 | 3 | 62
  Discharge up to 30 days: No Change | 12 | 61 | 118 | 116 | 23 | 7 | 337
  Discharge up to 30 days: Worsened 2 Classes | 0 | 1 | 2 | 1 | 0 | 0 | 4
  Discharge up to 30 days: Improved 2 Classes | 5 | 14 | 30 | 27 | 9 | 1 | 86
  Discharge up to 30 days: Improved 1 Class | 21 | 83 | 131 | 108 | 26 | 12 | 382
  Discharge up to 30 days: Worsened 3 Classes | 0 | 0 | 0 | 0 | 0 | 0 | 0
  3-6 Months: number analyzed (Participants) | 40 | 198 | 379 | 336 | 97 | 22 | 1073
  3-6 Months: Improved 3 Classes | 0 | 1 | 4 | 6 | 1 | 0 | 12
  3-6 Months: Improved 1 Class | 20 | 97 | 187 | 164 | 43 | 13 | 525
  3-6 Months: No Change | 5 | 47 | 76 | 79 | 25 | 4 | 236
  3-6 Months: Worsened 2 Classes | 0 | 0 | 0 | 0 | 0 | 0 | 0
  3-6 Months: Worsened 1 Class | 0 | 2 | 9 | 5 | 1 | 1 | 18
  3-6 Months: Improved 2 Classes | 15 | 51 | 103 | 82 | 27 | 4 | 282
  3-6 Months: Worsened 3 Classes | 0 | 0 | 0 | 0 | 0 | 0 | 0
  1 Year: number analyzed (Participants) | 37 | 196 | 369 | 322 | 93 | 17 | 1035
  1 Year: No Change | 8 | 47 | 76 | 70 | 26 | 3 | 230
  1 Year: Improved 1 Class | 16 | 83 | 176 | 161 | 40 | 10 | 486
  1 Year: Improved 3 Classes | 0 | 1 | 6 | 6 | 0 | 0 | 13
  1 Year: Improved 2 Classes | 13 | 60 | 105 | 79 | 27 | 4 | 289
  1 Year: Worsened 1 Class | 0 | 5 | 6 | 6 | 0 | 0 | 17
  1 Year: Worsened 2 Classes | 0 | 0 | 0 | 0 | 0 | 0 | 0
  1 Year: Worsened 3 Classes | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Effective Orifice Area Through 1 Year Post-procedure
Description: A minimum of 15 participants per valve size evaluated by transthoracic echocardiography technique and assessed by an independent core laboratory. The effective orifice area (EOA) is measured as the minimal cross-sectional area of the blood flow downstream of the aortic valve.
Time Frame: Discharge (up to 30 days), 3-6 months, 1 year post-implant
Population: At each timepoint, only subjects with echocardiography core lab data are included in the rows below.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Medtronic Avalus Valve 19mm | Medtronic Avalus Valve 21mm | Medtronic Avalus Valve 23mm | Medtronic Avalus Valve 25mm | Medtronic Avalus Valve 27mm | Medtronic Avalus Valve 29mm | Medtronic Avalus Valve (17mm - 29mm)
Number analyzed (Participants) | 42 | 211 | 401 | 350 | 101 | 26 | 1132
cm^2
  Discharge (up to 30 days): number analyzed (Participants) | 33 | 182 | 332 | 305 | 86 | 18 | 957
  Discharge (up to 30 days) | 1.23 (0.24) | 1.35 (0.30) | 1.59 (0.34) | 1.68 (0.37) | 1.88 (0.42) | 2.29 (0.68) | 1.60 (0.40)
  3-6 Months: number analyzed (Participants) | 40 | 181 | 356 | 319 | 90 | 19 | 1006
  3-6 Months | 1.22 (0.27) | 1.30 (0.26) | 1.54 (0.30) | 1.66 (0.32) | 1.89 (0.42) | 2.51 (0.71) | 1.57 (0.39)
  1 Year: number analyzed (Participants) | 34 | 184 | 352 | 312 | 86 | 17 | 986
  1 Year | 1.09 (0.23) | 1.26 (0.25) | 1.48 (0.33) | 1.60 (0.34) | 1.76 (0.35) | 2.42 (0.59) | 1.50 (0.38)

4. Primary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to the Effective Orifice Area Index (EOAI) Through 1 Year Post-implant
Description: A minimum of 15 participants per valve size evaluated by transthoracic echocardiography technique and assessed by an independent core laboratory for effective orifice area index (EOAI = EOA/BSA) Effective orifice area index is equal to the effective orifice area (EOA) in cm^2 divided by body surface area (BSA) in m^2.
  The achievement criterion for the effective orifice area index (EOAI) is defined to be ≥0.6 cm^2/m^2 12 months after the procedure. This criterion is in accordance with the definition of severe aortic stenosis in the American College of Cardiology (ACC) / American Heart Association (AHA) guidelines for the management of valvular heart disease.
Time Frame: Discharge (up to 30 days), 3-6 months, and 1 year post-implant
Population: At each timepoint, only subjects with echocardiography core lab data are included in the rows below.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Medtronic Avalus Valve 19mm | Medtronic Avalus Valve 21mm | Medtronic Avalus Valve 23mm | Medtronic Avalus Valve 25mm | Medtronic Avalus Valve 27mm | Medtronic Avalus Valve 29mm | Medtronic Avalus Valve (17mm - 29mm)
Number analyzed (Participants) | 42 | 211 | 401 | 350 | 101 | 26 | 1132
cm^2/m^2
  Discharge (up to 30 days): number analyzed (Participants) | 33 | 182 | 332 | 305 | 86 | 18 | 957
  Discharge (up to 30 days) | 0.71 (0.16) | 0.74 (0.18) | 0.81 (0.20) | 0.81 (0.19) | 0.89 (0.23) | 1.07 (0.3) | 0.81 (0.20)
  3-6 Months: number analyzed (Participants) | 40 | 181 | 356 | 319 | 90 | 19 | 1006
  3-6 Months | 0.71 (0.17) | 0.72 (0.16) | 0.79 (0.17) | 0.81 (0.17) | 0.90 (0.22) | 1.16 (0.31) | 0.80 (0.19)
  1 Year: number analyzed (Participants) | 34 | 184 | 352 | 312 | 86 | 17 | 986
  1 Year | 0.63 (0.14) | 0.70 (0.15) | 0.76 (0.18) | 0.78 (0.17) | 0.82 (0.17) | 1.14 (0.28) | 0.76 (0.18)

5. Primary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to the Peak Pressure Gradient (mmHg) From Discharge up to 1 Year
Description: A minimum of 15 participants per valve size evaluated by transthoracic echocardiography technique and assessed by an independent core laboratory.
  The peak pressure gradient is the maximum value measured of flow of blood through the aortic valve as measured in millimeters of mercury.
Time Frame: Measured at discharge (up to 30 days), 3-6 months, and 1 year post-implant
Population: At each timepoint, only subjects with echocardiography core lab data are included in the rows below.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Medtronic Avalus Valve 19mm | Medtronic Avalus Valve 21mm | Medtronic Avalus Valve 23mm | Medtronic Avalus Valve 25mm | Medtronic Avalus Valve 27mm | Medtronic Avalus Valve 29mm | Medtronic Avalus Valve (17mm - 29mm)
Number analyzed (Participants) | 42 | 211 | 401 | 350 | 101 | 26 | 1132
mmHg
  Discharge (up to 30 days): number analyzed (Participants) | 40 | 205 | 384 | 340 | 94 | 22 | 1086
  Discharge (up to 30 days) | 32.2 (9.7) | 28.0 (9.2) | 23.6 (8.0) | 22.4 (6.8) | 19.6 (6.8) | 16.2 (6.3) | 23.9 (8.4)
  3-6 Months: number analyzed (Participants) | 40 | 196 | 373 | 332 | 95 | 21 | 1058
  3-6 Months | 27.2 (6.7) | 26.3 (8.6) | 21.6 (6.8) | 21.1 (7.2) | 17.7 (5.9) | 14.7 (6.3) | 22.1 (7.7)
  1 Year: number analyzed (Participants) | 36 | 193 | 364 | 321 | 90 | 17 | 1022
  1 Year | 30.4 (8.2) | 27.8 (9.4) | 23.1 (7.5) | 22.0 (7.3) | 19.0 (6.7) | 18.1 (6.5) | 23.5 (8.3)

6. Primary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Mean Pressure Gradient (mmHg) Through 1 Year Post-implant
Description: A minimum of 15 participants per valve size evaluated by transthoracic echocardiography technique and will be assessed by an independent core laboratory. The mean pressure gradient is the average flow of blood through the aortic valve measured in millimeters of mercury.
Time Frame: Discharge (up to 30 days), 3-6 months, and 1 year post-implant
Population: At each timepoint, only subjects with echocardiography core lab data are included in the rows below.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Medtronic Avalus Valve 19mm | Medtronic Avalus Valve 21mm | Medtronic Avalus Valve 23mm | Medtronic Avalus Valve 25mm | Medtronic Avalus Valve 27mm | Medtronic Avalus Valve 29mm | Medtronic Avalus Valve (17mm - 29mm)
Number analyzed (Participants) | 42 | 211 | 401 | 350 | 101 | 26 | 1132
mmHg
  Discharge (up to 30 days): number analyzed (Participants) | 40 | 205 | 384 | 339 | 94 | 22 | 1085
  Discharge (up to 30 days) | 18.2 (6.1) | 15.2 (4.9) | 12.9 (4.5) | 12.4 (3.9) | 10.7 (3.8) | 8.8 (3.5) | 13.1 (4.7)
  3-6 Months: number analyzed (Participants) | 40 | 196 | 373 | 332 | 95 | 21 | 1058
  3-6 Months | 15.4 (4.4) | 14.2 (4.6) | 11.7 (3.7) | 11.3 (3.7) | 9.6 (3.3) | 7.9 (3.6) | 11.9 (4.1)
  1 Year: number analyzed (Participants) | 36 | 193 | 364 | 320 | 90 | 17 | 1021
  1 Year | 17.1 (5.0) | 15.1 (5.3) | 12.3 (4.0) | 11.9 (4.0) | 10.1 (3.7) | 10.2 (3.5) | 12.7 (4.6)

7. Primary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Performance Index (L/Min) Through 1 Year Post-implant
Description: A minimum of 15 participants per valve size will have performance index (L/Min) measured by transthoracic echocardiography technique and will be assessed by an independent core laboratory. The performance index is the measurement of the effective orifice area divided by the native orifice area.
Time Frame: Discharge (up to 30 days), 3-6 months, and 1 year post-implant
Population: At each timepoint, only subjects with echocardiography core lab data are included in the rows below.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Medtronic Avalus Valve 19mm | Medtronic Avalus Valve 21mm | Medtronic Avalus Valve 23mm | Medtronic Avalus Valve 25mm | Medtronic Avalus Valve 27mm | Medtronic Avalus Valve 29mm | Medtronic Avalus Valve (17mm - 29mm)
Number analyzed (Participants) | 42 | 211 | 401 | 350 | 101 | 26 | 1132
L/min
  Discharge (up to 30 days): number analyzed (Participants) | 33 | 182 | 332 | 305 | 86 | 18 | 957
  Discharge (up to 30 days) | 0.5 (0.1) | 0.5 (0.1) | 0.4 (0.1) | 0.4 (0.1) | 0.4 (0.1) | 0.4 (0.1) | 0.4 (0.1)
  3-6 Months: number analyzed (Participants) | 40 | 181 | 356 | 319 | 90 | 19 | 1006
  3-6 Months | 0.5 (0.1) | 0.4 (0.1) | 0.4 (0.1) | 0.4 (0.1) | 0.4 (0.1) | 0.4 (0.1) | 0.4 (0.1)
  1 Year: number analyzed (Participants) | 34 | 184 | 352 | 312 | 86 | 17 | 986
  1 Year | 0.5 (0.1) | 0.4 (0.1) | 0.4 (0.1) | 0.4 (0.1) | 0.3 (0.1) | 0.4 (0.1) | 0.4 (0.1)

8. Primary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Cardiac Output (L/Min) Through 1 Year Post-implant
Description: Cardiac output is the amount of blood pumped by the heart per minute. A minimum of 15 participants per valve size were evaluated for this outcome measure by transthoracic echocardiography technique and assessed by an independent core laboratory.
Time Frame: Discharge (up to 30 days), 3-6 months, and 1 year post-implant
Population: At each timepoint, only subjects with echocardiography core lab data are included in the rows below.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Medtronic Avalus Valve 19mm | Medtronic Avalus Valve 21mm | Medtronic Avalus Valve 23mm | Medtronic Avalus Valve 25mm | Medtronic Avalus Valve 27mm | Medtronic Avalus Valve 29mm | Medtronic Avalus Valve (17mm - 29mm)
Number analyzed (Participants) | 42 | 211 | 401 | 350 | 101 | 26 | 1132
L/min
  Discharge (up to 30 days): number analyzed (Participants) | 33 | 182 | 336 | 307 | 87 | 20 | 966
  Discharge (up to 30 days) | 5.0 (1.0) | 4.9 (1.2) | 5.1 (1.3) | 5.2 (1.2) | 5.3 (1.4) | 5.2 (1.2) | 5.1 (1.3)
  3-6 Months: number analyzed (Participants) | 40 | 180 | 357 | 319 | 90 | 19 | 1006
  3-6 Months | 4.6 (1.1) | 4.5 (0.9) | 4.8 (1.0) | 4.9 (1.1) | 4.9 (1.2) | 5.8 (1.7) | 4.8 (1.1)
  1 Year: number analyzed (Participants) | 34 | 186 | 351 | 313 | 86 | 17 | 988
  1 Year | 4.3 (1.0) | 4.5 (1.1) | 4.7 (1.1) | 4.9 (1.2) | 4.8 (1.0) | 6.4 (2.0) | 4.7 (1.2)

9. Primary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Cardiac Index (L/Min/m^2) Through 1 Year Post-implant
Description: A minimum of 15 participants per valve size evaluated by transthoracic echocardiography technique and will be assessed by an independent core laboratory.
  The cardiac index is an assessment of the cardiac output based on a patient's size measured by dividing the cardiac output by the patient's body's surface area.
Time Frame: Discharge (up to 30 days), 3-6 months, and 1 year post-implant
Population: At each timepoint, only subjects with echocardiography core lab data are included in the rows below.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Medtronic Avalus Valve 19mm | Medtronic Avalus Valve 21mm | Medtronic Avalus Valve 23mm | Medtronic Avalus Valve 25mm | Medtronic Avalus Valve 27mm | Medtronic Avalus Valve 29mm | Medtronic Avalus Valve (17mm - 29mm)
Number analyzed (Participants) | 42 | 211 | 401 | 350 | 101 | 26 | 1132
L/min/m^2
  Discharge (up to 30 days): number analyzed (Participants) | 33 | 182 | 336 | 307 | 87 | 20 | 966
  Discharge (up to 30 days) | 2.9 (0.7) | 2.7 (0.7) | 2.6 (0.7) | 2.5 (0.6) | 2.5 (0.7) | 2.4 (0.6) | 2.6 (0.7)
  3-6 Months: number analyzed (Participants) | 40 | 180 | 357 | 319 | 90 | 19 | 1006
  3-6 Months | 2.7 (0.7) | 2.5 (0.5) | 2.4 (0.5) | 2.4 (0.5) | 2.3 (0.6) | 2.7 (0.7) | 2.4 (0.5)
  1 Year: number analyzed (Participants) | 34 | 186 | 351 | 313 | 86 | 17 | 988
  1 Year | 2.5 (0.5) | 2.5 (0.6) | 2.4 (0.5) | 2.4 (0.6) | 2.2 (0.4) | 3.0 (0.8) | 2.4 (0.6)

10. Secondary Outcome: Evaluate the Safety of the Model 400 Avalus Valve With Regard to Valve-related Adverse Events and Death Annually Through 5 Years Post-implant
Description: Safety of the valve is evaluated by the time-related incidence of valve-related adverse events and death. The following valve-related adverse events are evaluated in this study: Thromboembolism, Thrombosis, Hemorrhage, Paravalvular leak (PVL), Endocarditis, Hemolysis, Structural valve deterioration, Non-structural dysfunction, Reintervention, Explant, and Death. The Kaplan-Meier event rates will be used to summarize valve-related adverse events and death. The Kaplan-Meier rate and the corresponding 95% confidence interval will be presented for each visit interval.
Time Frame: Annually, at years 2, 3, 4, and 5 post-implant
Reporting Status: Not Posted

11. Secondary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to the Change of New York Heart Association (NYHA) Classification From Baseline Through 5 Years Post-implant
Description: At each timepoint, participants were evaluated for change in New York Heart Association (NYHA) functional classification from baseline through 5 years post-procedure.
  Measure Description: Cardiac Disease with Functional Classes (lower value is more desirable than higher value) I - No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  II - Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  III - Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  IV - Symptoms of heart failure at rest. Any physical activity causes further discomfort.
Time Frame: Annually, at years 2, 3, 4, and 5 post-implant
Reporting Status: Not Posted

12. Secondary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Effective Orifice Area Through 5 Years Post-procedure
Description: Evaluated by transthoracic echocardiography technique and assessed by an independent core laboratory. The effective orifice area (EOA) is measured as the minimal cross-sectional area of the blood flow downstream of the aortic valve.
Time Frame: Annually, at years 2, 3, 4, and 5 post-implant
Reporting Status: Not Posted

13. Secondary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to the Effective Orifice Area Index (EOAI) Through 5 Years Post-implant
Description: Evaluated by transthoracic echocardiography technique and assessed by an independent core laboratory for effective orifice area index (EOAI = EOA/BSA) Effective orifice area index is equal to the effective orifice area (EOA) in cm^2 divided by body surface area (BSA) in m^2.
  The achievement criterion for the effective orifice area index (EOAI) is defined to be ≥0.6 cm^2/m^2 12 months after the procedure. This criterion is in accordance with the definition of severe aortic stenosis in the American College of Cardiology (ACC) / American Heart Association (AHA) guidelines for the management of valvular heart disease.
Time Frame: Annually, at years 2, 3, 4, and 5 post-implant
Reporting Status: Not Posted

14. Secondary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to the Peak Pressure Gradient (mmHg) From Discharge up to 5 Years Post-implant
Description: Evaluated by transthoracic echocardiography technique and assessed by an independent core laboratory.
  The peak pressure gradient is the maximum value measured of flow of blood through the aortic valve as measured in millimeters of mercury.
Time Frame: Annually, at years 2, 3, 4, and 5 post-implant
Reporting Status: Not Posted

15. Secondary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Mean Pressure Gradient (mmHg) Through 5 Years Post-implant
Description: Evaluated by transthoracic echocardiography technique and will be assessed by an independent core laboratory. The mean pressure gradient is the average flow of blood through the aortic valve measured in millimeters of mercury.
Time Frame: Annually, at years 2, 3, 4, and 5 post-implant
Reporting Status: Not Posted

16. Secondary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Performance Index (L/Min) Through 5 Years Post-implant
Description: Performance index (L/Min) measured by transthoracic echocardiography technique and will be assessed by an independent core laboratory. The performance index is the measurement of the effective orifice area divided by the native orifice area.
Time Frame: Annually, at years 2, 3, 4, and 5 post-implant
Reporting Status: Not Posted

17. Secondary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Cardiac Output (L/Min) Through 5 Years Post-implant
Description: Cardiac output is the amount of blood pumped by the heart per minute, evaluated by transthoracic echocardiography technique and assessed by an independent core laboratory.
Time Frame: Annually, at years 2, 3, 4, and 5 post-implant
Reporting Status: Not Posted

18. Secondary Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Cardiac Index (L/Min/m^2) Through 5 Years Post-implant
Description: Evaluated by transthoracic echocardiography technique and will be assessed by an independent core laboratory.
  The cardiac index is an assessment of the cardiac output based on a patient's size measured by dividing the cardiac output by the patient's body's surface area.
Time Frame: Annually, at years 2, 3, 4, and 5 post-implant
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Evaluate the Safety of the Model 400 Avalus Valve With Regard to Valve-related Adverse Events and Death at 1 Year Post-implant (Remaining Data From 29mm Valve Participants Not Required for Meeting Primary Outcomes)
Description: Safety of the valve is evaluated by the time-related incidence of valve-related adverse events and death. The following valve-related adverse events are evaluated in this study: Thromboembolism, Thrombosis, Hemorrhage, Paravalvular leak (PVL), Endocarditis, Hemolysis, Structural valve deterioration, Non-structural dysfunction, Reintervention, Explant, and Death. A minimum of 15 participants per valve size are evaluated. The Kaplan-Meier event rates will be used to summarize valve-related adverse events and death. The Kaplan-Meier rate and the corresponding 95% confidence interval will be presented for each visit interval.
Time Frame: 1 year post-implant
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to the Change of New York Heart Association (NYHA) Classification From Baseline Through 1 Year (Remaining Data From 29mm Valve Participants Not Required for Meeting Primary Outcomes)
Description: Participants evaluated for change in New York Heart Association (NYHA) functional classification from baseline to 1 year post-procedure.
  Measure Description: Cardiac Disease with Functional Classes (lower value is more desirable than higher value) I - No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  II - Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  III - Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  IV - Symptoms of heart failure at rest. Any physical activity causes further discomfort.
Time Frame: 3-6 months and 1 year post-implant
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Effective Orifice Area Through 1 Year Post-procedure (Remaining Data From 29mm Valve Participants Not Required for Meeting Primary Outcomes)
Description: as for outcome 12
Time Frame: 3-6 months, 1 year post-implant
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to the Effective Orifice Area Index (EOAI) Through 1 Year Post-implant (Remaining Data From 29mm Valve Participants Not Required for Meeting Primary Outcomes)
Description: as for outcome 13
Time Frame: 3-6 months, and 1 year post-implant
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to the Peak Pressure Gradient (mmHg) From Discharge up to 1 Year (Remaining Data From 29mm Valve Participants Not Required for Meeting Primary Outcomes)
Description: as for outcome 14
Time Frame: 3-6 months, and 1 year post-implant
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Mean Pressure Gradient (mmHg) Through 1 Year Post-implant (Remaining Data From 29mm Valve Participants Not Required for Meeting Primary Outcomes)
Description: as for outcome 15
Time Frame: 3-6 months, and 1 year post-implant
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Performance Index (L/Min) Through 1 Year Post-implant (Remaining Data From 29mm Valve Participants Not Required for Meeting Primary Outcomes)
Description: as for outcome 16
Time Frame: 3-6 months, and 1 year post-implant
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Cardiac Output (L/Min) Through 1 Year Post-implant (Remaining Data From 29mm Valve Participants Not Required for Meeting Primary Outcomes)
Description: Cardiac output is the amount of blood pumped by the heart per minute. Evaluated by transthoracic echocardiography technique and assessed by an independent core laboratory.
Time Frame: 3-6 months, and 1 year post-implant
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Cardiac Index (L/Min/m^2) Through 1 Year Post-implant (Remaining Data From 29mm Valve Participants Not Required for Meeting Primary Outcomes)
Description: as for outcome 18
Time Frame: 3-6 months, and 1 year post-implant
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve by Clinically Acceptable Hemodynamic Performance From Years 6 Through 12 Post-implant.
Description: Long-term follow-up clinically acceptable hemodynamic performance defined as freedom from surgical explant and/or percutaneous valve-in-valve reintervention due to structural valve deterioration
Time Frame: Annually, years 6-12 post-implant
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve From Years 6 - 12 Post-implant by Freedom From Valve-related Death
Time Frame: Annually, years 6 though 12 post-implant
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve From Years 6 - 12 Post-implant by Freedom From All-cause Mortality
Description: For time-to-event outcomes, Kaplan-Meier (actuarial) analysis of the event-free rate performed annually through twelve years.
Time Frame: Annually, years 6 though 12 post-implant
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve From Years 6 - 12 Post-implant by Change in NYHA Functional Classification Status From Baseline
Time Frame: Annually, years 6 though 12 post-implant
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Effective Orifice Area Through 12 Years Post-procedure
Description: as for outcome 12
Time Frame: Annually, years 6 though 12 post-implant
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to the Effective Orifice Area Index (EOAI) Through 12 Years Post-implant
Description: as for outcome 13
Time Frame: Annually, years 6 though 12 post-implant
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to the Peak Pressure Gradient (mmHg) up to 12 Years Post-implant
Description: as for outcome 14
Time Frame: Annually, years 6 though 12 post-implant
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Mean Pressure Gradient (mmHg) Through 12 Years Post-implant
Description: as for outcome 15
Time Frame: Annually, years 6 though 12 post-implant
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Performance Index (L/Min) Through 12 Years Post-implant
Description: as for outcome 16
Time Frame: Annually, years 6 though 12 post-implant
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Cardiac Output (L/Min) Through 12 Years Post-implant
Description: as for outcome 26
Time Frame: Annually, years 6 though 12 post-implant
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Confirm the Effectiveness of the Model 400 Avalus Valve With Regard to Cardiac Index (L/Min/m^2) Through 12 Years Post-implant
Description: as for outcome 18
Time Frame: Annually, years 6 though 12 post-implant
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Site reported adverse events and serious adverse events data collected from implant through 1 year.
Description: Site reported events for a minimum of 15 subjects per valve size through 1 year post-implant.
Groups:
- Medtronic Avalus Valve (All valve sizes): All participants implanted with the with Medtronic Avalus Valve (sized 17mm - 29mm) from procedure through 1 year.
Arm/Group | Medtronic Avalus Valve (All valve sizes)
All-Cause Mortality (participants affected / at risk) | 170/1132
Serious Adverse Events (participants affected / at risk) | 638/1132
Other Adverse Events (participants affected / at risk) | 1105/1132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic Avalus Valve (All valve sizes) (N=1132)
Anaemias Haemolytic Immune (Blood And Lymphatic System Disorders) | 1 (1)
Anaemias Nec (Blood And Lymphatic System Disorders) | 98 (106)
Bleeding Tendencies (Blood And Lymphatic System Disorders) | 2 (2)
Coagulopathies (Blood And Lymphatic System Disorders) | 10 (10)
Haemolyses Nec (Blood And Lymphatic System Disorders) | 1 (1)
Leukocytoses Nec (Blood And Lymphatic System Disorders) | 2 (2)
Leukopenias Nec (Blood And Lymphatic System Disorders) | 1 (1)
Spleen Disorders (Blood And Lymphatic System Disorders) | 1 (1)
Thrombocytopenias (Blood And Lymphatic System Disorders) | 18 (18)
Cardiac Conduction Disorders (Cardiac Disorders) | 49 (55)
Cardiac Disorders Nec (Cardiac Disorders) | 5 (5)
Cardiomyopathies (Cardiac Disorders) | 2 (2)
Coronary Artery Disorders Nec (Cardiac Disorders) | 12 (12)
Heart Failures Nec (Cardiac Disorders) | 43 (46)
Ischaemic Coronary Artery Disorders (Cardiac Disorders) | 13 (13)
Left Ventricular Failures (Cardiac Disorders) | 2 (2)
Mitral Valvular Disorders (Cardiac Disorders) | 6 (6)
Myocardial Disorders Nec (Cardiac Disorders) | 5 (5)
Noninfectious Pericarditis (Cardiac Disorders) | 6 (6)
Pericardial Disorders Nec (Cardiac Disorders) | 49 (54)
Rate And Rhythm Disorders Nec (Cardiac Disorders) | 5 (5)
Supraventricular Arrhythmias (Cardiac Disorders) | 146 (167)
Tricuspid Valvular Disorders (Cardiac Disorders) | 1 (1)
Ventricular Arrhythmias And Cardiac Arrest (Cardiac Disorders) | 31 (31)
Cardiac Septal Defects Congenital (Congenital, Familial And Genetic Disorders) | 1 (1)
Inner Ear Signs And Symptoms (Ear And Labyrinth Disorders) | 1 (1)
Thyroid Disorders Nec (Endocrine Disorders) | 1 (1)
Optic Nerve Bleeding And Vascular Disorders (Eye Disorders) | 2 (2)
Retinal Structural Change, Deposit And Degeneration (Eye Disorders) | 1 (1)
Visual Impairment And Blindness (Excl Colour Blindness) (Eye Disorders) | 1 (1)
Acute And Chronic Pancreatitis (Gastrointestinal Disorders) | 2 (2)
Anal And Rectal Disorders Nec (Gastrointestinal Disorders) | 1 (1)
Anal And Rectal Ulcers And Perforation (Gastrointestinal Disorders) | 1 (1)
Benign Neoplasms Gastrointestinal (Excl Oral Cavity) (Gastrointestinal Disorders) | 4 (4)
Colitis (Excl Infective) (Gastrointestinal Disorders) | 1 (1)
Diaphragmatic Hernias (Gastrointestinal Disorders) | 2 (2)
Diarrhoea (Excl Infective) (Gastrointestinal Disorders) | 1 (1)
Diverticula (Gastrointestinal Disorders) | 2 (2)
Duodenal And Small Intestinal Stenosis And Obstruction (Gastrointestinal Disorders) | 1 (1)
Duodenal Ulcers And Perforation (Gastrointestinal Disorders) | 5 (5)
Gastric And Oesophageal Haemorrhages (Gastrointestinal Disorders) | 2 (2)
Gastritis (Excl Infective) (Gastrointestinal Disorders) | 1 (1)
Gastrointestinal Atonic And Hypomotility Disorders Nec (Gastrointestinal Disorders) | 2 (2)
Gastrointestinal Signs And Symptoms Nec (Gastrointestinal Disorders) | 2 (2)
Gastrointestinal Stenosis And Obstruction Nec (Gastrointestinal Disorders) | 3 (3)
Gastrointestinal Ulcers And Perforation, Site Unspecified (Gastrointestinal Disorders) | 1 (1)
Gastrointestinal Vascular Occlusion And Infarction (Gastrointestinal Disorders) | 1 (1)
Inguinal Hernias (Gastrointestinal Disorders) | 4 (4)
Intestinal Haemorrhages (Gastrointestinal Disorders) | 7 (7)
Non-Mechanical Ileus (Gastrointestinal Disorders) | 1 (1)
Non-Site Specific Gastrointestinal Haemorrhages (Gastrointestinal Disorders) | 11 (11)
Peritoneal And Retroperitoneal Disorders (Gastrointestinal Disorders) | 1 (1)
Cardiac Complications Associated With Device (General Disorders And Administration Site Conditions) | 8 (9)
Complications Associated With Device Nec (General Disorders And Administration Site Conditions) | 3 (3)
Death And Sudden Death (General Disorders And Administration Site Conditions) | 1 (1)
Febrile Disorders (General Disorders And Administration Site Conditions) | 6 (6)
General Signs And Symptoms Nec (General Disorders And Administration Site Conditions) | 9 (9)
Healing Abnormal Nec (General Disorders And Administration Site Conditions) | 5 (5)
Hernias Nec (General Disorders And Administration Site Conditions) | 1 (1)
Oedema Nec (General Disorders And Administration Site Conditions) | 2 (2)
Pain And Discomfort Nec (General Disorders And Administration Site Conditions) | 3 (3)
Vascular Complications Associated With Device (General Disorders And Administration Site Conditions) | 1 (1)
Cholecystitis And Cholelithiasis (Hepatobiliary Disorders) | 7 (7)
Cholestasis And Jaundice (Hepatobiliary Disorders) | 1 (1)
Hepatic And Hepatobiliary Disorders Nec (Hepatobiliary Disorders) | 2 (2)
Hepatic Failure And Associated Disorders (Hepatobiliary Disorders) | 2 (2)
Obstructive Bile Duct Disorders (Excl Neoplasms) (Hepatobiliary Disorders) | 1 (1)
Structural And Other Bile Duct Disorders (Hepatobiliary Disorders) | 1 (1)
Allergies To Foods, Food Additives, Drugs And Other Chemicals (Immune System Disorders) | 4 (4)
Anaphylactic And Anaphylactoid Responses (Immune System Disorders) | 4 (4)
Abdominal And Gastrointestinal Infections (Infections And Infestations) | 3 (3)
Bacterial Infections Nec (Infections And Infestations) | 9 (9)
Bone And Joint Infections (Infections And Infestations) | 1 (1)
Cardiac Infections (Infections And Infestations) | 15 (16)
Clostridia Infections (Infections And Infestations) | 1 (1)
Coronavirus Infections (Infections And Infestations) | 1 (1)
Fungal Infections Nec (Infections And Infestations) | 2 (2)
Herpes Viral Infections (Infections And Infestations) | 1 (1)
Infections Nec (Infections And Infestations) | 16 (19)
Lower Respiratory Tract And Lung Infections (Infections And Infestations) | 36 (39)
Sepsis, Bacteraemia, Viraemia And Fungaemia Nec (Infections And Infestations) | 31 (33)
Streptococcal Infections (Infections And Infestations) | 1 (1)
Upper Respiratory Tract Infections (Infections And Infestations) | 2 (2)
Urinary Tract Infections (Infections And Infestations) | 9 (11)
Vascular Infections (Infections And Infestations) | 1 (1)
Viral Infections Nec (Infections And Infestations) | 2 (2)
Abdominal And Gastrointestinal Injuries Nec (Injury, Poisoning And Procedural Complications) | 1 (1)
Anaesthetic And Allied Procedural Complications (Injury, Poisoning And Procedural Complications) | 1 (1)
Bone And Joint Injuries Nec (Injury, Poisoning And Procedural Complications) | 1 (1)
Cardiac And Vascular Procedural Complications (Injury, Poisoning And Procedural Complications) | 15 (15)
Cardiovascular Injuries (Injury, Poisoning And Procedural Complications) | 5 (5)
Cerebral Injuries Nec (Injury, Poisoning And Procedural Complications) | 1 (1)
Eye Injuries Nec (Injury, Poisoning And Procedural Complications) | 1 (1)
Gastrointestinal And Hepatobiliary Procedural Complications (Injury, Poisoning And Procedural Complications) | 1 (1)
Limb Fractures And Dislocations (Injury, Poisoning And Procedural Complications) | 2 (2)
Medication Errors, Product Use Errors And Issues Nec (Injury, Poisoning And Procedural Complications) | 1 (1)
Nerve Injuries Nec (Injury, Poisoning And Procedural Complications) | 1 (1)
Non-Site Specific Injuries Nec (Injury, Poisoning And Procedural Complications) | 2 (2)
Non-Site Specific Procedural Complications (Injury, Poisoning And Procedural Complications) | 55 (57)
Respiratory Tract And Thoracic Cavity Procedural Complications (Injury, Poisoning And Procedural Complications) | 8 (10)
Site Specific Injuries Nec (Injury, Poisoning And Procedural Complications) | 2 (2)
Skin Injuries Nec (Injury, Poisoning And Procedural Complications) | 2 (2)
Spinal Fractures And Dislocations (Injury, Poisoning And Procedural Complications) | 1 (1)
Thoracic Cage Fractures And Dislocations (Injury, Poisoning And Procedural Complications) | 1 (1)
Urinary Tract Procedural Complications (Injury, Poisoning And Procedural Complications) | 1 (1)
Carbohydrate Tolerance Analyses (Incl Diabetes) (Investigations) | 1 (1)
Cardiac Function Diagnostic Procedures (Investigations) | 3 (3)
Coagulation And Bleeding Analyses (Investigations) | 1 (1)
Mineral And Electrolyte Analyses (Investigations) | 1 (1)
Protein Analyses Nec (Investigations) | 1 (1)
Red Blood Cell Analyses (Investigations) | 3 (3)
Renal Function Analyses (Investigations) | 1 (1)
Respiratory Tract And Thoracic Histopathology Procedures (Investigations) | 1 (1)
Skeletal And Cardiac Muscle Analyses (Investigations) | 1 (1)
Vascular Tests Nec (Incl Blood Pressure) (Investigations) | 1 (1)
White Blood Cell Analyses (Investigations) | 1 (1)
Disorders Of Purine Metabolism (Metabolism And Nutrition Disorders) | 2 (2)
Hyperglycaemic Conditions Nec (Metabolism And Nutrition Disorders) | 4 (4)
Metabolic Acidoses (Excl Diabetic Acidoses) (Metabolism And Nutrition Disorders) | 3 (3)
Sodium Imbalance (Metabolism And Nutrition Disorders) | 3 (3)
Total Fluid Volume Decreased (Metabolism And Nutrition Disorders) | 4 (4)
Total Fluid Volume Increased (Metabolism And Nutrition Disorders) | 4 (5)
Cartilage Disorders (Musculoskeletal And Connective Tissue Disorders) | 1 (1)
Joint Related Disorders Nec (Musculoskeletal And Connective Tissue Disorders) | 1 (1)
Muscle Weakness Conditions (Musculoskeletal And Connective Tissue Disorders) | 1 (1)
Musculoskeletal And Connective Tissue Conditions Nec (Musculoskeletal And Connective Tissue Disorders) | 1 (1)
Musculoskeletal And Connective Tissue Pain And Discomfort (Musculoskeletal And Connective Tissue Disorders) | 12 (12)
Myopathies (Musculoskeletal And Connective Tissue Disorders) | 1 (2)
Osteoarthropathies (Musculoskeletal And Connective Tissue Disorders) | 7 (7)
Spine And Neck Deformities (Musculoskeletal And Connective Tissue Disorders) | 2 (2)
Bladder Neoplasms Malignant (Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps)) | 1 (1)
Breast And Nipple Neoplasms Malignant (Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps)) | 1 (1)
Central Nervous System Neoplasms Malignant Nec (Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps)) | 1 (1)
Endocrine Neoplasms Malignant And Unspecified Nec (Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps)) | 1 (1)
Female Reproductive Neoplasms Unspecified Malignancy (Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps)) | 1 (1)
Gallbladder Neoplasms Malignant (Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps)) | 1 (1)
Laryngeal Neoplasms Malignant (Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps)) | 1 (1)
Leukaemias Acute Myeloid (Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps)) | 1 (1)
Lower Gastrointestinal Neoplasms Benign (Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps)) | 1 (1)
Myelodysplastic Syndromes (Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps)) | 1 (1)
Neoplasms Malignant Site Unspecified Nec (Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps)) | 21 (21)
Prostatic Neoplasms Malignant (Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps)) | 1 (1)
Renal Neoplasms Benign (Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps)) | 1 (1)
Renal Neoplasms Malignant (Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps)) | 1 (1)
Urinary Tract Neoplasms Unspecified Malignancy Nec (Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps)) | 2 (2)
Acute Polyneuropathies (Nervous System Disorders) | 1 (1)
Central Nervous System Haemorrhages And Cerebrovascular Accidents (Nervous System Disorders) | 37 (38)
Central Nervous System Vascular Disorders Nec (Nervous System Disorders) | 3 (3)
Coordination And Balance Disturbances (Nervous System Disorders) | 1 (1)
Dementia (Excl Alzheimer's Type) (Nervous System Disorders) | 1 (1)
Disturbances In Consciousness Nec (Nervous System Disorders) | 10 (11)
Encephalopathies Nec (Nervous System Disorders) | 3 (3)
Encephalopathies Toxic And Metabolic (Nervous System Disorders) | 2 (2)
Headaches Nec (Nervous System Disorders) | 1 (1)
Hydrocephalic Conditions (Nervous System Disorders) | 1 (1)
Increased Intracranial Pressure Disorders (Nervous System Disorders) | 1 (1)
Lumbar Spinal Cord And Nerve Root Disorders (Nervous System Disorders) | 2 (2)
Neurological Signs And Symptoms Nec (Nervous System Disorders) | 4 (4)
Neuromuscular Disorders Nec (Nervous System Disorders) | 1 (1)
Parkinson's Disease And Parkinsonism (Nervous System Disorders) | 1 (1)
Peripheral Neuropathies Nec (Nervous System Disorders) | 1 (1)
Seizures And Seizure Disorders Nec (Nervous System Disorders) | 9 (9)
Spinal Cord And Nerve Root Disorders Nec (Nervous System Disorders) | 2 (2)
Structural Brain Disorders Nec (Nervous System Disorders) | 1 (1)
Transient Cerebrovascular Events (Nervous System Disorders) | 14 (14)
Tremor (Excl Congenital) (Nervous System Disorders) | 2 (2)
Device Incompatibility Issues (Product Issues) | 3 (3)
Device Issues Nec (Product Issues) | 2 (2)
Device Malfunction Events Nec (Product Issues) | 1 (1)
Anxiety Symptoms (Psychiatric Disorders) | 1 (1)
Confusion And Disorientation (Psychiatric Disorders) | 12 (12)
Delusional Symptoms (Psychiatric Disorders) | 1 (1)
Depressive Disorders (Psychiatric Disorders) | 1 (1)
Mental Disorders Nec (Psychiatric Disorders) | 9 (9)
Substance Related And Addictive Disorders (Psychiatric Disorders) | 2 (2)
Bladder And Urethral Symptoms (Renal And Urinary Disorders) | 6 (6)
Nephritis Nec (Renal And Urinary Disorders) | 1 (1)
Renal Disorders Nec (Renal And Urinary Disorders) | 1 (1)
Renal Failure And Impairment (Renal And Urinary Disorders) | 38 (45)
Renal Lithiasis (Renal And Urinary Disorders) | 3 (4)
Renal Obstructive Disorders (Renal And Urinary Disorders) | 1 (1)
Urinary Abnormalities (Renal And Urinary Disorders) | 1 (1)
Testicular And Epididymal Disorders Nec (Reproductive System And Breast Disorders) | 1 (1)
Breathing Abnormalities (Respiratory, Thoracic And Mediastinal Disorders) | 9 (9)
Bronchospasm And Obstruction (Respiratory, Thoracic And Mediastinal Disorders) | 2 (2)
Conditions Associated With Abnormal Gas Exchange (Respiratory, Thoracic And Mediastinal Disorders) | 5 (5)
Coughing And Associated Symptoms (Respiratory, Thoracic And Mediastinal Disorders) | 3 (3)
Lower Respiratory Tract Inflammatory And Immunologic Conditions (Respiratory, Thoracic And Mediastinal Disorders) | 1 (1)
Lower Respiratory Tract Signs And Symptoms (Respiratory, Thoracic And Mediastinal Disorders) | 1 (1)
Mediastinal Disorders (Respiratory, Thoracic And Mediastinal Disorders) | 10 (10)
Nasal Disorders Nec (Respiratory, Thoracic And Mediastinal Disorders) | 1 (1)
Parenchymal Lung Disorders Nec (Respiratory, Thoracic And Mediastinal Disorders) | 3 (3)
Pneumothorax And Pleural Effusions Nec (Respiratory, Thoracic And Mediastinal Disorders) | 111 (119)
Pulmonary Oedemas (Respiratory, Thoracic And Mediastinal Disorders) | 11 (11)
Pulmonary Thrombotic And Embolic Conditions (Respiratory, Thoracic And Mediastinal Disorders) | 6 (6)
Respiratory Failures (Excl Neonatal) (Respiratory, Thoracic And Mediastinal Disorders) | 40 (43)
Respiratory Tract Disorders Nec (Respiratory, Thoracic And Mediastinal Disorders) | 3 (3)
Dermal And Epidermal Conditions Nec (Skin And Subcutaneous Tissue Disorders) | 1 (1)
Rashes, Eruptions And Exanthems Nec (Skin And Subcutaneous Tissue Disorders) | 1 (1)
Skin Injuries And Mechanical Dermatoses (Skin And Subcutaneous Tissue Disorders) | 1 (1)
Skin Preneoplastic Conditions Nec (Skin And Subcutaneous Tissue Disorders) | 1 (1)
Cardiac Device Therapeutic Procedures (Surgical And Medical Procedures) | 1 (1)
Cardiac Therapeutic Procedures Nec (Surgical And Medical Procedures) | 1 (1)
Gastrointestinal Therapeutic Procedures Nec (Surgical And Medical Procedures) | 1 (1)
Therapeutic Procedures Nec (Surgical And Medical Procedures) | 1 (1)
Aortic Aneurysms And Dissections (Vascular Disorders) | 4 (4)
Aortic Necrosis And Vascular Insufficiency (Vascular Disorders) | 4 (4)
Circulatory Collapse And Shock (Vascular Disorders) | 1 (1)
Haemorrhages Nec (Vascular Disorders) | 2 (2)
Lymphangiopathies (Vascular Disorders) | 2 (2)
Non-Site Specific Embolism And Thrombosis (Vascular Disorders) | 4 (4)
Non-Site Specific Necrosis And Vascular Insufficiency Nec (Vascular Disorders) | 1 (1)
Non-Site Specific Vascular Disorders Nec (Vascular Disorders) | 1 (1)
Peripheral Embolism And Thrombosis (Vascular Disorders) | 3 (4)
Peripheral Vascular Disorders Nec (Vascular Disorders) | 2 (2)
Site Specific Necrosis And Vascular Insufficiency Nec (Vascular Disorders) | 1 (1)
Site Specific Vascular Disorders Nec (Vascular Disorders) | 6 (6)
Vascular Hypertensive Disorders Nec (Vascular Disorders) | 9 (9)
Vascular Hypotensive Disorders (Vascular Disorders) | 26 (26)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic Avalus Valve (All valve sizes) (N=1132)
Anaemias Nec (Blood And Lymphatic System Disorders) | 420 (446)
Leukocytoses Nec (Blood And Lymphatic System Disorders) | 87 (89)
Thrombocytopenias (Blood And Lymphatic System Disorders) | 255 (267)
Cardiac Conduction Disorders (Cardiac Disorders) | 396 (532)
Heart Failures Nec (Cardiac Disorders) | 69 (85)
Pericardial Disorders Nec (Cardiac Disorders) | 167 (184)
Supraventricular Arrhythmias (Cardiac Disorders) | 674 (930)
Tricuspid Valvular Disorders (Cardiac Disorders) | 77 (79)
Ventricular Arrhythmias And Cardiac Arrest (Cardiac Disorders) | 128 (139)
Gastrointestinal Atonic And Hypomotility Disorders Nec (Gastrointestinal Disorders) | 65 (68)
Nausea And Vomiting Symptoms (Gastrointestinal Disorders) | 96 (104)
Oedema Nec (General Disorders And Administration Site Conditions) | 183 (189)
Lower Respiratory Tract And Lung Infections (Infections And Infestations) | 73 (85)
Urinary Tract Infections (Infections And Infestations) | 70 (76)
Gastrointestinal And Hepatobiliary Procedural Complications (Injury, Poisoning And Procedural Complications) | 58 (61)
Non-Site Specific Procedural Complications (Injury, Poisoning And Procedural Complications) | 276 (328)
Physical Examination Procedures And Organ System Status (Investigations) | 73 (73)
Electrolyte Imbalance Nec (Metabolism And Nutrition Disorders) | 70 (75)
Hyperglycaemic Conditions Nec (Metabolism And Nutrition Disorders) | 220 (231)
Potassium Imbalance (Metabolism And Nutrition Disorders) | 60 (67)
Total Fluid Volume Increased (Metabolism And Nutrition Disorders) | 65 (66)
Musculoskeletal And Connective Tissue Pain And Discomfort (Musculoskeletal And Connective Tissue Disorders) | 127 (138)
Neurological Signs And Symptoms Nec (Nervous System Disorders) | 83 (86)
Confusion And Disorientation (Psychiatric Disorders) | 120 (126)
Bladder And Urethral Symptoms (Renal And Urinary Disorders) | 101 (110)
Renal Failure And Impairment (Renal And Urinary Disorders) | 164 (186)
Breathing Abnormalities (Respiratory, Thoracic And Mediastinal Disorders) | 77 (80)
Parenchymal Lung Disorders Nec (Respiratory, Thoracic And Mediastinal Disorders) | 127 (133)
Pneumothorax And Pleural Effusions Nec (Respiratory, Thoracic And Mediastinal Disorders) | 387 (442)
Pulmonary Oedemas (Respiratory, Thoracic And Mediastinal Disorders) | 122 (125)
Respiratory Failures (Excl Neonatal) (Respiratory, Thoracic And Mediastinal Disorders) | 129 (138)
Vascular Hypertensive Disorders Nec (Vascular Disorders) | 158 (184)
Vascular Hypotensive Disorders (Vascular Disorders) | 225 (252)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 60 days of receipt Medtronic (MDT) will verify presence of Confidential Information (CI) & won't censor or interfere with presentation/conclusions except to protect CI (other than Study Data) & its rights in patentable or copyrightable materials, & check technical accuracy of MDT data. If told by MDT that Publication contains CI or technical errors of MDT data, PI will make requested changes before publishing/presenting. PI will delay publication up to 90 more days, if requested.

DOCUMENTS (3):
  • Study Protocol (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT02088554/Prot_003.pdf
  • Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT02088554/SAP_004.pdf
  • Informed Consent Form (2015-03-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT02088554/ICF_002.pdf